CLINICAL TRIAL: NCT03198247
Title: Physiotherapy and Therapeutic Education in Patients With Pain Catastrophizing After a Total Knee Arthroplasty. Randomized Clinical Trial
Brief Title: Physiotherapy and Therapeutic Education After Total Knee Arthroplasty.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low participation
Sponsor: Centro Universitario La Salle (Other)
Collaborators: Hospital Clinic of Barcelona (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Hector Beltran-Alacreu, PhD, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKA-01
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — galactosylceramide sulfotransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Usual Care (Active Comparator): Procedure: Usual care The biomedical education session will be imparted 2 weeks before surgery by the preoperative nurse and a physiotherapist. It will have a duration of 2 hours and it is designed for a group of 5 subjects.
  The hospital rehabilitation starts 6 hours after surgery, and it is based in early wandering stimulation, articular mobility exercises and isometric exercises.
  Interventions: Other: Usual care
- Experimental: Usual Care + PNE and CST (Experimental): Procedure: Usual care + PNE and CST. The PNE and CST program will be divided in 3 individual sessions. This program is mainly based in "Explain Pain" concept, used in multiple rehabilitation programs. Its aim is to change the subject's pain understanding, teaching them the biological processes underneath the pain construct, as a mechanism to reduce itself and its related maladaptative thoughts and behaviours
  Interventions: Other: Usual care; Other: PNE + CST

INTERVENTIONS:
Other: Usual care — The biomedical education session will be imparted 2 weeks before surgery by the preoperative nurse and a physiotherapist. It will have a duration of 2 hours and it is designed for a group of 5 subjects.
  The hospital rehabilitation starts 6 hours after surgery, and it is based in early wandering stimulation, articular mobility exercises and isometric exercises.
Other: PNE + CST — The PNE and CST program will be divided in 3 individual sessions.
  Arms: Experimental: Usual Care + PNE and CST

SUMMARY:
The purpose of this study is to test whether adding a treatment using pain neuroscience education (PNE) and coping skills training (CST) to usual care, in subjects with knee osteoarthritis and pain catastrophizing, who are scheduled for a total knee arthroplasty (TKA), is more effective than only usual care. There is a high evidence level of different systematic reviews, which support the efficacy of physiotherapy treatments combined with behavioural techniques aimed to reduce pain catastrophism, pain and disability in other pathologies. The primary aim of that kind of interventions is to help the subjects to reconceptualise its own pain understanding and its role on the recovery process, as well as promoting an increase of activity and encourage the subject to resume its usual activity instead of continuing to avoid it.

DETAILED DESCRIPTION:
The prevalence of TKA has increased dramatically during the last two decades, its popularity can be attributed to its evident success regarding pain improvement, deformity correction and disability reduction in knee osteoarthritis subjects. However, only a third of the patients report no functional problems after surgery, the 20% of then are unsatisfied with its functional skills and around a 20% are experiencing pain, high disability degrees and a significant quality of life reduction. This results cannot be fully explained by mechanical processes, surgical procedures or surgery variations, but it seems to be related to other psychological aspects. Chronic pain subjects often develop maladaptative thoughts and behaviours (i.e. pain catastrophism, Kinesiophobia, activity avoidance) which contribute to make the subject suffer physically as well as emotionally, and affect on the intensity and persistency of pain.

Although many psychosocial factors have been studied, pain catastrophism has emerged as one of the most important predictors for persistent pain after a total knee arthroplasty, as well as its severity and duration, that's why it is getting more importance when it comes to study chronic pain in this subjects. Reducing pain catastrophism has become a key factor to determine the success in the rehabilitation of some maladies accompanied by pain, considering that its reduction has been associated with the clinical improvement of pain itself. It has been observed that treatments using psychological and psychosocial interventions, therapeutic education and coping skills training, or physical therapy and therapeutic exercise, are effective techniques to reduce pain catastrophism. Nevertheless, it's still necessary to determine whether the maladaptative pain related thoughts approach, using physical therapy and behavioural techniques, are able to reduce the risk of suffering postoperative chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. To have sufficient Spanish or Catalan reading, writing and speaking skills to comprehend all explanations and to complete the assessment tools.
2. Be able to provide the informed consent.
3. Be scheduled to undergo in a total knee arthroplasty.
4. Knee osteoarthritis diagnosis.
5. Score more than 16 points in the PCS.
6. Patients between 65-80 years.

Exclusion Criteria:

1. Patients scheduled to undergo in a total knee arthroplasty because of prostheses replacement, tumor, infection or fracture.
2. Patients scheduled to undergo in a bilateral total knee arthroplasty.
3. Patients that will need another total knee or hip replacement surgery in less than a year regarding the current intervention.
4. Patients scheduled for unicompartmental knee arthroplasty.
5. Patients with other pathologies with characteristic features of a central sensitization. (i.e. Fibromyalgia)
6. Co-existing other inflammatory or rheumatic conditions (i.e. rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus or ankylosing spondylitis)
7. Co-existing other mental condition and/or major depression.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life. Changes from Baseline to 6 months | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete the Euro Quality of Life (QoL) Score (EQ-5D) (Spanish version),

SECONDARY OUTCOMES:
Disability / limitations | Baseline, 3 and 6 months after surgical intervention
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC) (Spanish version) will be used to assess patient´s physical function. This questionnaire can be completed in less than 5 minutes. It's a widely used, reliable, valid and responsive measure of outcome in people with osteoarthritis of the hip or knee.
Pain intensity | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to rate their pain on a horizontal 100-mm Visual Analogue Scale (VAS). The horizontal line anchors will be "no pain" and "worst imaginable pain". The VAS is a valid and reliable instrument compared with other pain rating scales, and has been well established in clinical practice and research for measuring pain levels in arthritis populations.
Function | Baseline, 3 and 6 months after surgical intervention
  30-Second Chair Stand Test will be use to evaluate patient's functionality on standing, because it is a well-recognized test to detect early declines in functional independence.
Range of Motion | Baseline, 3 and 6 months after surgical intervention
  Goniometric assessments of knee will be carried out to assess flexion and extension range of motion.
Neuropathic Pain | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete Self-Administered Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) (Spanish version).
Pain Catastrophizing | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete the Pain Catastrophizing Scale (PCS) (Spanish version).
Kinesiophobia | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete the Tampa Scale for Kinesiophobia (TSK-11) (Spanish version).
Self-efficacy | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete the Chronic Pain Self-Efficacy Scale (Spanish version).
Self-coping ability | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete the "Cuestionario de Afrontamiento ante el Dolor Crónico - Versión Reducida" (CAD-R)), a Spanish questionnaire to asses self-coping ability.
Depression and anxiety | Baseline, 3 and 6 months after surgical intervention
  Participants will be asked to complete the Hospital Anxiety and Depression Scale (HADS) (Spanish version) will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, España, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ochandorena-Acha M, Escriba-Salvans A, Hernandez-Hermoso JA, Terradas-Monllor M. Perioperative experiences of patients with high pain catastrophizing and knee arthroplasty after receiving or not preoperative physiotherapy: Qualitative study. Musculoskelet Sci Pract. 2024 Apr;70:102918. doi: 10.1016/j.msksp.2024.102918. Epub 2024 Feb 2. PMID 38330866